CLINICAL TRIAL: NCT04633317
Title: Aerosolized Colistin to Mechanical Ventilated Patients With CRGNB Pneumonia
Brief Title: Aerosolized Colistin to Mechanical Ventilated Patients With Pneumonia
Acronym: CRGNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Ling Lin, Associate professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRPD1K0861
Record Dates: First submitted 2020-11-14; First posted 2020-11-18 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia, Bacterial
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Regimen (Experimental): Randomized 80 subjects diagnosed with pneumonia of carbapenem-resistant gram negative bacteria will received inhaled colistimethate sodium generated by a pneumatic nebulizer or a vibrating mesh nebulizer every 12 hours for 7-10 days
  Interventions: Device: A pneumatic nebulizer; Device: A vibrating mesh nebulizer
- Group B Regimen (No Intervention): Randomized 40 subjects diagnosed with pneumonia of carbapenem-resistant gram negative bacteria will received inhaled colistimethate sodium intravenous every 12 hours for 7-10 days

INTERVENTIONS:
Device: A pneumatic nebulizer — Inhaled colistimethate sodium generated by a pneumatic nebulizer
  Arms: Group A Regimen
Device: A vibrating mesh nebulizer — Inhaled colistimethate sodium generated by a vibrating mesh nebulizer
  Arms: Group A Regimen

SUMMARY:
The purpose of this study was to determine the effect of aerosolized colistin on to ventilated patients with carbapenem-resistant gram negative bacteria pneumonia. We hypothesize that adjunct aerosolized colistin, which achieve high drug concentrations in the airway, would more effectively treat the penumbra.

DETAILED DESCRIPTION:
To treat respiratory infection of patients with mechanical ventilation, greater systemic antibiotic dose is required through the patient's venous injection. In this trial, patients with arbapenem-resistant gram negative bacteria pneumonia (CRGNB)were assigned to adjunct aerosolized colistin delivered by a jet nebulizer or a vibrating mesh nebulizer comparing to or standard intravenous injection by a randomizing protocol.

Need for a systemic antibiotic was determined by the clinical physician. Comparisons were made between standard care and study drug for their effects on bacteria eradiation, incidence of nephrotoxicity, and oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Patients received invasive mechanical ventilation >48 hours
* Diagnosed with pneumonia caused by carbapenem resistance gram negative bacteria

Exclusion Criteria:

* pregnant or lactating women
* receiving colistin > 3 days
* recurrent pneumonia caused by carbapenem resistance gram negative bacteria
* allergy to colistin or polymyxin B drugs
* immunocompromised, defined as neutropenia ANC<500 cells/ul
* HIV positive
* received chemotherapy with 3 months
* renal function deficiency (creatinine clearance < 30 ml/min)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical pulmonary infection score | 7-10 days
  The clinical pulmonary infection score calculated on the basis of points assigned for various signs and symptoms of pneumonia (eg, fever and extent of oxygenation impairment

SECONDARY OUTCOMES:
Ventilator pressure control level | 7-10 days
  Ventilator pressure control level setting indirectly indicate lung compliance

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, MS, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Huang CC, Fang TP, Lin CM, Chu CM, Hsiao HL, Liu JF, Li HH, Chiu LC, Kao KC, Kuo CH, Leu SW, Lin HL. Evaluating the Efficacy of Inhaled Colistin via Two Nebulizer Types in Ventilator-Associated Pneumonia: Prospective Randomized Trial. Antibiotics (Basel). 2024 Nov 19;13(11):1099. doi: 10.3390/antibiotics13111099. PMID 39596792